CLINICAL TRIAL: NCT05760690
Title: Single-center, Retrospective Study of Retro-Auricular Single-Site Endoscopic, Transoral Endoscopic Thyroidectomy Vestibular Approach and Transareola Endoscopic Thyroidectomy in Patients With Early Stage Papillary Thyroid Carcinoma
Brief Title: Safety of Endoscopic Thyroidectomy Via Retro-Auricular Single-Site Approach, Transoral Approach and Transareola
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ouyang Dian, Clinical Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-359-01
Record Dates: First submitted 2023-02-13; First posted 2023-03-08 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: Papillary Thyroid Carcinoma Laparoscopy; Endoscopic Thyroidectomy; Retroauricular Single-site approach; Transoral Endoscopic Thyroidectomy Vestibular Approach; Transareola Endoscopic Thyroidectomy
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Retro-Auricular Single-Site Endoscopic Thyroidectomy group (Experimental): Patients in the retro-auricular single-site endoscopic thyroidectomy (RASSET) group will receive endoscopic thyroid lobectomy and central lymph node dissection.
  Interventions: Procedure: Retro-Auricular Single-Site Endoscopic Thyroidectomy
- Transoral Endoscopic Thyroidectomy Vestibular Approach group (Active Comparator): Patients in the Transoral Endoscopic Thyroidectomy Vestibular Approach group will receive endoscopic thyroid lobectomy and central lymph node dissection.
  Interventions: Procedure: Transoral Endoscopic Thyroidectomy Vestibular Approach
- Transareola Endoscopic Thyroidectomy group (Active Comparator): Patients in the Transareola Endoscopic Thyroidectomy group will receive endoscopic thyroid lobectomy and central lymph node dissection.
  Interventions: Procedure: Transareola Endoscopic Thyroidectomy

INTERVENTIONS:
Procedure: Retro-Auricular Single-Site Endoscopic Thyroidectomy — The strap muscles and the sternocleidomastoid muscle were separated. Upper parathyroid and lower parathyroid glands were identified and preserved. The recurrent laryngeal nerve (RLN) was identified，A lobe of thyroid specimen and central lymph nodes were dissected.
  Arms: Retro-Auricular Single-Site Endoscopic Thyroidectomy group
Procedure: Transoral Endoscopic Thyroidectomy Vestibular Approach — The patient was placed in a supine position with slight neck extension under nasotracheal intubation. The mouth was garbled with povidone iodine before surgery. Three laparoscopic ports (a 10- to 15-mm port at midline and two 5-mm ports at the lateral junction between the canine and first premolar teeth)were inserted under the lower lip at the oral vestibular area.The strap muscleswere separated in the midline to expose the thyroid and trachea. The recurrent laryngeal nerve (RLN) was identified at the insertion to the larynx, then followed downandparallel tothe trachea inferiorly.
  Arms: Transoral Endoscopic Thyroidectomy Vestibular Approach group
Procedure: Transareola Endoscopic Thyroidectomy — The patient was in supine position. Incision was made inside the right areola and a 10mm puncture device was placed, subcutaneous separation rod was used to separate the space, and a 30° endoscope was introduced, puncture device was placed in a 5mm incision on the left areola, ultrasonic knife free flap was used, subcutaneous separation space was placed in the upper sternal segment, and a 5mm puncture device was placed outside the right areola. The anterior cervical flap was further dissociated to establish a space. The median cervical line was cut to cut off the isthmus of the thyroid, and the tracheal fascia ligament of the thyroid was separated and the nerve was exposed to protect the nerves. Then remove the lobe of thyroid and central lymph nodes
  Arms: Transareola Endoscopic Thyroidectomy group

SUMMARY:
The goal of this retrospective study is to compare the safety and efficiacy of endoscopic thyroidectomy via retro-auricular single-site approach, transoral endoscopic thyroidectomy vestibular approach and transareola approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, no gender restrictions.
2. Fine-needle aspiration cytology(FNA) confirmed papillary thyroid carcinoma(PTC).
3. Early stage PTC (stage T1N0M0).
4. Preoperative ultrasonography showed unilateral glandular lobe malignant tumor and the largest diameter was not more than 2cm, without cervical lymph node metastasis and extensive metastasis.
5. Patients undergoing thyroid lobectomy and central lymph node dissection.
6. Patients who have signed an approved Informed Consent.

Exclusion Criteria:

1. Patients who do not accept case data collection for various reasons.
2. The clinical data unfit this study (at the discretion of the investigator).
3. Patients who have undergone neck surgery or radiotherapy before this trail.
4. Patients who have uncontrolled hyperthyroidism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
C-reactive protein，CRP | 1 week
  the level of CRP before and after operation

SECONDARY OUTCOMES:
Serum Amyloid A，SAA | 1 week
  the level of CRP before and after operation
blood loss | 1 week
  The volume of blood loss during operation
VAS pain score | 2 days after operation
  Postoperative VAS score was recorded
number of lymph nodes | 1 week after operation
  Postoperative specimen Postoperative specimen Postoperative specimen Postoperative specimen the number of lymph nodes in postoperative specimens

CONTACTS AND LOCATIONS:
Overall Officials: Dian Ouyang, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong F, Yang A, Ouyang D. Retroauricular Single-Site Endoscopic Thyroidectomy-A Balanced Endoscopic Approach for Thyroid Excision. JAMA Surg. 2023 May 1;158(5):548-549. doi: 10.1001/jamasurg.2022.7723. PMID 36753130
- [Background] Dong F, Ao Y, Li MT, Zhan ZR, Lin YQ, Tan QJ, Li H, Yang AK, Ouyang D. [A comparative study between retro-auricular single-site endoscopic thyroidectomy and transoral endoscopic thyroidectomy vestibular approach: a single-center retrospective analysis]. Zhonghua Wai Ke Za Zhi. 2021 Nov 1;59(11):891-896. doi: 10.3760/cma.j.cn112139-20210903-00420. Chinese. PMID 34743449
- [Background] Liang TJ, Chen IS, Liu SI. Working Space Creation in Transoral Thyroidectomy: Pearls and Pitfalls. Cancers (Basel). 2022 Feb 17;14(4):1031. doi: 10.3390/cancers14041031. PMID 35205779
- [Background] Sun H, Zheng H, Wang X, Zeng Q, Wang P, Wang Y. Comparison of transoral endoscopic thyroidectomy vestibular approach, total endoscopic thyroidectomy via areola approach, and conventional open thyroidectomy: a retrospective analysis of safety, trauma, and feasibility of central neck dissection in the treatment of papillary thyroid carcinoma. Surg Endosc. 2020 Jan;34(1):268-274. doi: 10.1007/s00464-019-06762-6. Epub 2019 Jul 25. PMID 31346748
- [Background] Ikeda Y, Takami H, Niimi M, Kan S, Sasaki Y, Takayama J. Endoscopic thyroidectomy and parathyroidectomy by the axillary approach. A preliminary report. Surg Endosc. 2002 Jan;16(1):92-5. doi: 10.1007/s004640080175. Epub 2001 Nov 12. PMID 11961613
- [Background] Anuwong A, Ketwong K, Jitpratoom P, Sasanakietkul T, Duh QY. Safety and Outcomes of the Transoral Endoscopic Thyroidectomy Vestibular Approach. JAMA Surg. 2018 Jan 1;153(1):21-27. doi: 10.1001/jamasurg.2017.3366. PMID 28877292
- [Background] Russell JO, Razavi CR, Al Khadem MG, Lopez M, Saraf S, Prescott JD, Starmer HM, Richmon JD, Tufano RP. Anterior cervical incision-sparing thyroidectomy: Comparing retroauricular and transoral approaches. Laryngoscope Investig Otolaryngol. 2018 Sep 24;3(5):409-414. doi: 10.1002/lio2.200. eCollection 2018 Oct. PMID 30410996
- [Background] Sephton BM. Extracervical Approaches to Thyroid Surgery: Evolution and Review. Minim Invasive Surg. 2019 Aug 20;2019:5961690. doi: 10.1155/2019/5961690. eCollection 2019. PMID 31531238
- [Background] Lee DW, Ko SH, Song CM, Ji YB, Kim JK, Tae K. Comparison of postoperative cosmesis in transaxillary, postauricular facelift, and conventional transcervical thyroidectomy. Surg Endosc. 2020 Aug;34(8):3388-3397. doi: 10.1007/s00464-019-07113-1. Epub 2019 Sep 12. PMID 31515625

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT05760690/Prot_SAP_000.pdf